CLINICAL TRIAL: NCT05400395
Title: A Prospective, Randomized, Placebo-controlled, Double-blinded, Multi-center, Phase IV, Exploratory Clinical Trial to Demonstrate the Effect of Improving the Walking Distance by GNX80 in Patients With Intermittent Claudication
Brief Title: Clinical Trial for GNX80 in Intermittent Claudication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNX_001
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNX (Experimental): GNX / 80mg / BID / PO
  Interventions: Drug: GNX80
- Placebo (Placebo Comparator): Placebo / BID / PO
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GNX80 — GNX80 oral intake(BID) for 24 weeks
  Other Names: Test
  Arms: GNX
Drug: Placebo — Placebo oral intake(BID) for 24 weeks
  Other Names: Control
  Arms: Placebo

SUMMARY:
This is a Phase 4, randomized clinical trial to evaluate whether GNX80 vs. placebo, prescribed for 6 months to patients with Intermittent Claudication(IC) would lead to an improvement in the walking distance.

DETAILED DESCRIPTION:
A Prospective, Randomized, Placebo-controlled, Double-blinded, Multi-center, Phase IV, Exploratory Clinical Trial to Demonstrate the Effect of Improving the Walking Distance by GNX80 in Patients with Intermittent Claudication

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 20 years
* Angiographically confirmed peripheral arterial disease
* Intermittent claudication for more than 6 months

Exclusion Criteria:

* Severe impairment of heart, liver, or kidney function
* Limitation of walking ability due to respiratory insufficiency or to an orthopaedic condition
* Poorly controlled diabetes mellitus
* Positive pregnancy test
* Planned surgical or endovascular procedures other than for the treatment of IC

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Walking Distance in comparison with the findings from at baseline | 24 weeks
  walking distance evaluated by a constant treadmill test

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea